CLINICAL TRIAL: NCT07325812
Title: Effect of Periodic Alveolar Recruitment Maneuvers on Intraoperative Atelectasis and Dynamic Respiratory Mechanics Assessed by Lung Ultrasound in Adult Patients Undergoing Elective Lumbar Spine Surgery in the Prone Position: A Randomized Controlled Trial
Brief Title: Effect of Periodic Alveolar Recruitment Maneuvers on Intraoperative Atelectasis in Adult Patients Undergoing Prone Lumbar Spine Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, SERAP KARACALAR, Professor of Anesthesiology and Reanimation, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CTERHO-SOZER-LUS-ARM-PRONE-001
Record Dates: First submitted 2025-12-25; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Atelectasis; Mechanical Ventilation; General Anesthesia; Prone Position
Keywords: Atelectasis; Alveolar Recruitment Maneuver; Lung Ultrasound; Prone Position; Respiratory Mechanics
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 1:1 ratio to one of two parallel groups. All participants will receive a standardized baseline alveolar recruitment maneuver after prone positioning. In the intervention group, additional alveolar recruitment maneuvers will be applied at regular intervals during surgery, while participants in the control group will not receive further recruitment maneuvers beyond the baseline intervention. Participants will remain in their assigned group for the duration of the study.
Who Masked: Outcomes Assessor
Masking Description: Lung ultrasound examinations and outcome assessments will be performed by an investigator who is blinded to group allocation. The anesthesiology team providing intraoperative care and performing the recruitment maneuvers will not be blinded due to the nature of the intervention. Participants will be under general anesthesia and therefore will not be aware of group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Periodic Alveolar Recruitment Maneuver Group (Experimental): Participants assigned to this arm will receive standard general anesthesia and mechanical ventilation. After placement in the prone position, a baseline ultrasound-guided alveolar recruitment maneuver will be performed in all participants. In this arm, additional alveolar recruitment maneuvers will be applied at regular intervals during surgery, approximately once every hour, in order to maintain lung aeration throughout the procedure.
  Interventions: Procedure: Alveolar Recruitment Maneuver
- Single Baseline Alveolar Recruitment Maneuver Group (Active Comparator): Participants assigned to this arm will receive standard general anesthesia and mechanical ventilation. After placement in the prone position, a single baseline ultrasound-guided alveolar recruitment maneuver will be performed. No additional alveolar recruitment maneuvers will be applied during the remainder of the surgical procedure, and ventilation will otherwise follow standard intraoperative management.
  Interventions: Procedure: Alveolar Recruitment Maneuver

INTERVENTIONS:
Procedure: Alveolar Recruitment Maneuver — An alveolar recruitment maneuver will be applied under general anesthesia using a closed ventilatory system. Following prone positioning, a baseline recruitment maneuver will be performed by applying continuous positive airway pressure of approximately 30-40 cmH₂O for 5-10 seconds. Depending on group assignment, the recruitment maneuver will either be repeated at regular intraoperative intervals (approximately once every hour) or applied only once as a single baseline maneuver.
  Other Names: Lung Recruitment Maneuver

SUMMARY:
During general anesthesia, especially when patients are placed in the prone (face-down) position for spine surgery, parts of the lungs may partially collapse. This condition, called atelectasis, can reduce oxygen levels and affect breathing during and after surgery. Although anesthesiologists routinely use a breathing technique known as an alveolar recruitment maneuver to reopen collapsed lung areas, performing this maneuver only once at the beginning of surgery may not be sufficient to keep the lungs open throughout longer procedures.

The purpose of this study is to determine whether performing alveolar recruitment maneuvers at regular intervals during surgery can better prevent lung collapse compared with performing a single maneuver at the start of surgery. The study will include adult patients undergoing elective lumbar spine surgery under general anesthesia in the prone position.

All participants will receive standard anesthesia care and a baseline alveolar recruitment maneuver after being positioned for surgery. Participants will then be randomly assigned to one of two groups. One group will receive additional alveolar recruitment maneuvers approximately once every hour during surgery, while the other group will not receive further recruitment maneuvers beyond the initial one. Lung aeration will be assessed using lung ultrasound, a non-invasive imaging method that does not involve radiation.

The main outcome of the study is the presence of significant lung collapse immediately before removal of the breathing tube at the end of surgery. Secondary outcomes include measurements of breathing mechanics, oxygen levels, and the occurrence of temporary drops in oxygen saturation. The results of this study may help determine the most effective way to maintain lung function during prone spine surgery and improve respiratory safety during anesthesia.

DETAILED DESCRIPTION:
Detailed Description

General anesthesia and mechanical ventilation are known to reduce functional residual capacity and promote the development of atelectasis, particularly during prolonged surgical procedures. The prone position, which is commonly required for lumbar spine surgery, may further exacerbate these effects by altering chest wall mechanics and increasing intraabdominal and intrathoracic pressures. Intraoperative atelectasis has been associated with impaired oxygenation and adverse respiratory outcomes in the perioperative period.

Alveolar recruitment maneuvers are routinely used in anesthetic practice to reopen collapsed lung units and improve lung aeration. However, evidence from pediatric populations suggests that a single recruitment maneuver followed by standard positive end-expiratory pressure may be insufficient to maintain lung aeration during prolonged prone positioning. Whether a strategy of repeated, periodic recruitment maneuvers provides additional benefit in adult patients undergoing prone spine surgery remains unclear.

This prospective, single-center, randomized controlled trial is designed to evaluate the effect of periodic intraoperative alveolar recruitment maneuvers on lung aeration and respiratory mechanics in adult patients undergoing elective lumbar spine surgery in the prone position. After induction of standardized general anesthesia and placement of the patient in the prone position, lung aeration will be assessed using lung ultrasound. Lung ultrasound is a bedside, radiation-free imaging modality that allows regional evaluation of lung aeration and detection of atelectasis through validated scoring systems.

All participants will receive a baseline ultrasound-guided alveolar recruitment maneuver after the initial lung ultrasound assessment in the prone position. Following this baseline intervention, participants will be randomized to one of two parallel groups. In the periodic recruitment group, alveolar recruitment maneuvers will be repeated at regular intervals during surgery, approximately once per hour. In the control group, no additional recruitment maneuvers will be performed beyond the initial baseline maneuver. Ventilation settings and anesthetic management will otherwise be standardized and consistent between groups.

Lung ultrasound examinations will be performed at predefined intraoperative time points by an investigator who is blinded to group allocation. Lung aeration will be quantified using a standardized lung ultrasound scoring approach, allowing comparison of the incidence and severity of atelectasis between groups. In addition to lung ultrasound findings, intraoperative respiratory mechanics, including peak inspiratory pressure and dynamic lung compliance, will be recorded at predefined time points. Oxygen saturation will be monitored continuously, and episodes of oxygen desaturation will be documented.

The primary objective of the study is to compare the incidence of significant intraoperative atelectasis between patients receiving periodic alveolar recruitment maneuvers and those receiving a single baseline maneuver. Secondary objectives include evaluation of differences in respiratory mechanics, oxygenation parameters, and the occurrence of transient intraoperative or early postoperative respiratory events. Safety outcomes related to recruitment maneuvers, such as transient hypotension or oxygen desaturation, will also be monitored.

By assessing lung aeration with lung ultrasound and focusing on a practical ventilation strategy that can be easily implemented during routine anesthesia care, this study aims to provide clinically relevant data on optimizing intraoperative respiratory management in adult patients undergoing prone lumbar spine surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 65 years

Scheduled for elective lumbar spine surgery under general anesthesia

Surgery planned to be performed in the prone position

Expected surgical duration of at least 90 minutes

American Society of Anesthesiologists (ASA) physical status I-II

Ability to provide written informed consent

Exclusion Criteria:

* Body mass index (BMI) greater than 30 kg/m²

History of thoracic surgery

Known or suspected chronic pulmonary disease (e.g., chronic obstructive pulmonary disease, restrictive lung disease)

Clinically significant cardiac disease

Pregnancy or breastfeeding

Known airway anomalies

Intraoperative conversion to a surgical duration shorter than 90 minutes

Refusal or inability to provide informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of Significant Intraoperative Atelectasis Assessed by Lung Ultrasound | Immediately before tracheal extubation at the end of surgery
  Significant intraoperative atelectasis will be defined as the presence of lung consolidation detected by lung ultrasound, corresponding to a lung ultrasound aeration score of 2 or higher in at least one predefined lung region. Lung ultrasound examinations will be performed using a standardized scanning protocol, and images will be evaluated by an outcome assessor blinded to group allocation.

SECONDARY OUTCOMES:
Peak Inspiratory Pressure | Intraoperatively, at predefined time points during surgery
  Peak inspiratory pressure will be recorded during mechanical ventilation as an indicator of airway pressure and respiratory system mechanics. Measurements will be obtained using the anesthesia ventilator at predefined intraoperative time points.
Dynamic Lung Compliance | Intraoperatively, at predefined time points during surgery
  Dynamic lung compliance will be calculated from ventilator-derived measurements as an indicator of respiratory system compliance during mechanical ventilation. Values will be recorded at predefined intraoperative time points.
Peripheral Oxygen Saturation | Intraoperatively and during early postoperative recovery (up to 30 minutes in the post-anesthesia care unit)
  Peripheral oxygen saturation will be continuously monitored using standard pulse oximetry. Recorded values will be used to assess intraoperative and early postoperative oxygenation status.
Incidence of Oxygen Desaturation | Intraoperatively and during early postoperative recovery (up to 30 minutes in the post-anesthesia care unit)
  Oxygen desaturation will be defined as a peripheral oxygen saturation value below 95% recorded during intraoperative monitoring or early postoperative recovery.